CLINICAL TRIAL: NCT04578236
Title: Efficacy of Aerosol Combination Therapy of 13 Cis Retinoic Acid and Captopril for Treating Covid-19 Patients Via Indirect Inhibition of Transmembrane Protease, Serine 2 (TMPRSS2)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Faculty of Science, Damietta University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARS
Record Dates: First submitted 2020-10-04; First posted 2020-10-08 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerosolized 13 cis retinoic acid plus Inhalation administration by nebulization captopril 25mg (Experimental): Infected patients will receive aerosolized 13 cis retinoic acid in gradual one dose per day increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days plus Inhalation administration by nebulization captopril 25mg for 14 days
  Interventions: Combination Product: Aerosolized 13 cis retinoic acid plus Inhalation administration by nebulization captopril 25mg
- The standard therapy (Sham Comparator): infected patients will receive the standard therapy for COVID-19 for 14 days
  Interventions: Drug: Drug: Standard treatment Standard treatment

INTERVENTIONS:
Combination Product: Aerosolized 13 cis retinoic acid plus Inhalation administration by nebulization captopril 25mg — Infected patients will receive aerosolized 13 cis retinoic acid in gradual one dose per day increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days plus Inhalation administration by nebulization captopril 25mg for 14 days
  Arms: Aerosolized 13 cis retinoic acid plus Inhalation administration by nebulization captopril 25mg
Drug: Drug: Standard treatment Standard treatment — Drug: Standard treatment Standard treatment is according to the protocol of treatment of 2019-nCoV infection
  Arms: The standard therapy

SUMMARY:
Efficacy of Aerosol Combination Therapy of 13 Cis Retinoic Acid and Captopril for Treating Covid-19 Patients Via Indirect Inhibition of Transmembrane Protease, Serine 2 (TMPRSS2)

Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) has infected over 20,000,000 people causing over 700,000 deaths. It has no currently approved treatments.Airborne SARS-CoV-2 infections in humans initiate from the virus entering nasal and airway epithelial cells through binding to angiotensin-converting enzyme 2 (ACE2). Transmembrane protease, serine 2 (TMPRSS2), a cellular protease that activates the SARS-CoV-2 spike protein, colocalizes with ACE2 and can prime SARS-CoV-2 fusion directly at the plasma membrane. Transmembrane protease, serine 2 (TMPRSS2) is an androgen receptor signaling target gene and an androgen-regulated cell-surface serine protease expressed predominantly in prostate and lung epithelial cell. TMPRSS2 is normally expressed several folds higher in the prostate relative to any other human tissue, though the normal physiological function(s) remains unknown. A study found that dihydrotestosterone (DHT) s a potent activator of TMPRSS2.On the other hand, Feily et al noted that low-dose isotretinoin (0.5 mg/kg/day for 15-20 weeks) in PCO patients with moderate to severe nodulocystic acne resulted in significant decreases in levels of serum total testosterone, prolactin, and dihydrotestosterone A study demonstrated that 13- cis -Retinoic acid competitively and reversibly inhibits dihydrotestosterone. Therefore, we suggest that 13- cis -Retinoic acid will downregulate TMPRSS2 expression thorough temporary preventing the effect of dihydrotestosterone (DHT) on the activation of TMPRSS2 gene expression. ACE inhibitors and ARBs are commonly taken by heart patients to reduce blood pressure and to treat heart failure.Earlier studies had cautioned that this class of drugs could possibly increase the risk for the novel coronavirus, SARS-CoV-2, infection and elevate COVID-19 severity. There is conflicting observational evidence about the potential clinical impact of ACE inhibitors and ARBs on patients with COVID-19. Select preclinical investigations have raised concerns about their safety in patients with COVID-19. On the other hand, Preliminary data hypothesise that angiotensin-converting enzyme (ACE) inhibitors and renin-angiotensin- aldosterone system (RAAS) inhibitors could benefit patients with COVID-19 by decreasing acute lung damage and preventing angiotensin-II-mediated pulmonary inflammation. Here in our review, we use established and emerging evidence based on the findings of previous studies and researches to propose that ACE inhibitors may benefit patients with COVID-19 via attenuating and abolishing the effect of androgenic hormones on inducing the expression of Transmembrane protease, serine 2 (TMPRSS2), even though, at the same time, ACE inhibitors cause an increase in the human cell surface receptor protein ACE2 which the novel coronavirus uses to enter and infect cells. A study on hypertensive rats demonstrated that using ACE inhibitors(captopril) abolished and attenuated the effect of dihydrotestosterone (DHT). In this study RAS inhibition exhibited beneficial effects on androgen-induced obesity and abolished the androgen-mediated increase in blood pressure (BP) observed in this model of PCOS. (83 ± 1 vs 115 ± 3 mmHg, p<0.0001). A another study found that the angiotensin converting enzyme inhibitor captopril abolished testosterone effect and attenuates testosterone-induced benign prostatic hyperplasia in rats; a mechanistic approach. Captopril is a potent inhibitor of the angiotensin converting enzyme. These effects of testosterone were almost prevented by captopril (100 mg/kg). In conclusion, generally treatment with ACE inhibitors is associated with reduced androgen levels. Therefore,we think that Transmembrane protease, serine 2 (TMPRSS2) is an indirect target of ACE inhibitors and 13 cis retinoic acid As aresult, we hypothesize that any drug which downregulates TMPRSS2 expression through targeting AR, AR co-regulatory factors, or AR downstream transcription factors might be potentially effective against COVID-19 and is worth investigating under a clinical trial..

Keywords: COVID -19, Transmembrane protease, serine 2 (TMPRSS2), ACE inhibitors, ACE2.

DETAILED DESCRIPTION:
This is a Phase 2, , randomized (1:1:1), placebo-controlled, 2-weeks, proof-of-concept study to evaluate the safety and tolerability as well as the mechanistic effect of Aerosol administration of Aerosolized 13 cis retinoic acid plus Inhalation administration by nebulization captopril 25mg in subjects infected with COVID -19

After randomization and standard treatment The infected patients will receive Aerosolized 13 cis retinoic acid plus Inhalation administration by nebulization captopril 25mg once daily. for 14 days

Outcome Measures

* Primary Outcome Measure
* lung injury score
* Proportion of lung injury score decreased or increased after treatmen [Time Frame: at 7and 14 days]

Secondary Outcome Measures:

* Transe membrane protease ,serine II (TMPRSS2) changes over time [Time Frame: at day 7 and 14]
* Testosterone levels changes over time [Time Frame: at day 7 and 14]
* Dihydrotestosterone(DHT) levels changes over time [Time Frame: at day 7 and 14]]
* Cholesterol levels changes over time [Time Frame: at day 7 and 14]
* Angiotensin 1-7 (Ang 1-7) changes over time [Time Frame: at day 7 and 14]
* Angiotensin 1-5 (Ang 1-5) changes over time [Time Frame: at day 7 and 14]
* Renin changes over time [Time Frame: at day 7 and 14]
* Aldosterone changes over time [Time Frame: at day 7 and 14]
* Angiotensin-converting enzyme (ACE) changes over time [Time Frame: at day 7 and 14]
* Time to first negative SARS-CoV-2 PCR in NP swap [Time Frame: day 7 and 14]
* All cause mortality rate [Time Frame: day 7 and 14]
* Ventilation free days [Time Frame: day 7 and 14]
* ICU free days [Time Frame: day 7 and 14]

ELIGIBILITY:
Inclusion Criteria:

Adult SARI patients with 2019-ncov infection confirmed by PCR; Absolute value of lymphocytes < 0. 6x 109/L; Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

Age < 18 Pregnant Allergic to experimental drugs and patients have the following conditions:

* Hypercholesterolemia
* Hypertriglyceridemia
* Liver disease
* Renal disease
* Sjögren syndrome
* Pregnancy
* Lactation
* Depressive disorder
* Body mass index less than 18 points or higher than 25 points
* Contraindications for hormonal contraception or intrauterine device.
* Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation
* Patients receiving anti-hcv treatment
* Permanent blindness in one eye
* History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery
* History of ACE-inhibitor allergy
* History of angio-oedema
* Co-infection with another respiratory pathogen which could be responsible of pneumonia
* Hypersensitivity to captopril, to any other angiotensin converting enzyme inhibitor or any of the excipients of the specialty used
* Shock requiring vasopressor infusion
* Patient on state medical ai
* The competent physician considered it inappropriate to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
lung injury score | at 7days
  Proportion of lung injury score decreased or increased after treatmen

SECONDARY OUTCOMES:
Transe membrane protease ,serine II (TMPRSS2) changes over time | at day 7 and 14
Testosterone levels changes over time | at day 7 and 14
Dihydrotestosterone(DHT) levels changes over time | at day 7 and 14]
Cholesterol levels changes over time | at day 7 and 14
Angiotensin 1-7 (Ang 1-7) changes over time | at day 7 and 14
Angiotensin 1-5 (Ang 1-5) changes over time | at day 7 and 14
Renin changes over time | at day 7 and 14
Aldosterone changes over time | at day 7 and 14
Angiotensin-converting enzyme (ACE) changes over time | at day 7 and 14
Time to first negative SARS-CoV-2 PCR in NP swap | day 7 and 14
All cause mortality rate | day 7 and 14
Ventilation free days | day 7 and 14
ICU free days | day 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Elkazzaz, B.Sc in Biochemistry, Principal Investigator — Faculty of Science, Damietta University

IPD SHARING:
Plan to Share IPD: No